CLINICAL TRIAL: NCT01462110
Title: Determination of Anti-Plaque and Anti-Gingivitis Efficacy of One Experimental Mouthrinse Following a Baseline Oral Prophylaxis: A Four Week Study
Brief Title: A Four-Week Study to Measure the Effectiveness of an Experimental Mouthwash Used After Teeth Cleaning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: LAEBBA0001
Record Dates: First submitted 2011-10-26; First posted 2011-10-31 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Dental Plaque
Keywords: Gingivitis; Microorganisms
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- 0.15% ethyl lauroyl arginate HCl-containing mouthrinse (Experimental): Brush teeth as usual, followed immediately by rinsing with 20 mL of assigned 0.15% ethyl lauroyl arginate HCl-containing mouthrinse (19415-154-1) for 30 seconds - repeat twice daily for four weeks.
  Interventions: Device: 19416-154-1
- 5% hydroalcohol mouthrinse (Sham Comparator): Brush teeth as usual, followed immediately by rinsing with 20 mL of assigned 5% hydroalcohol mouthrinse (W002194-0221P) for 30 seconds - repeat twice daily for four weeks.
  Interventions: Device: W002194-0221P

INTERVENTIONS:
Device: 19416-154-1 — 0.15% ethyl lauroyl arginate HCl-containing mouthrinse
  Other Names: Not Marketed
  Arms: 0.15% ethyl lauroyl arginate HCl-containing mouthrinse
Device: W002194-0221P — 5% hydroalcohol mouthrinse
  Other Names: Not Marketed
  Arms: 5% hydroalcohol mouthrinse

SUMMARY:
This study will test the idea that using an experimental mouth rinse after each time you brush your teeth will result in a healthier mouth than using the regular mouth rinse. Participants will be expected to avoid oral hygiene (like brushing teeth or using mouthwash) for at least 12 hours before each visit and will not be allowed to eat, drink or smoke for at least 4 hours before each visit.

At the first visit, the study will be explained to you in detail and you will be allowed to ask any questions you may have before signing a consent form. You will complete a medical/dental history and the dentist will examine your mouth, during which he will poke your gums and scrape some plaque off your teeth for testing. If you do not meet the requirements to continue in the trial, you will be told that you do not need to return for more testing.

If you meet requirements to continue, you will have an equal chance of being assigned to use either of the two mouth rinses being studied. You will be given a diary, toothbrush, toothpaste, and your assigned mouth rinse, with instructions on how they must be used.

You will be instructed not to use any unassigned oral care products and to follow your usual eating habits. You will be given appointments to return two times within the next four weeks. At those visits, the staff will check to make sure you're following the instructions and ask how you're feeling, and the dentist will do the same thing he did during the first visit.

DETAILED DESCRIPTION:
The primary objective of this randomized, double-blind, single-center, controlled, parallel-designed clinical study is to determine the efficacy of an experimental mouth rinse on whole-mouth mean plaque and gingivitis scores as an adjunct to brushing after four weeks of use.

The secondary objectives will be to determine the efficacy of the an experimental mouth rinse as an adjunct to brushing on whole-mouth mean plaque and gingivitis measured at 2 weeks as well as a bleeding assessment according to the Bleeding Index at 2 and 4 weeks. A microbiological assessment will be performed to identify and quantify specific oral microbes to assess any change in population.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age and in good general health.
* Must display adequate oral hygiene (i.e., brush teeth daily and exhibit no signs of oral neglect).
* Volunteers must read, sign, and receive a copy of the Informed Consent Form after the nature of the study has been fully explained.
* Must be willing to use the products according to instructions and be available for appointments.
* Baseline dental measurements meet protocol-specified criteria.
* Willingness to refrain from using all oral hygiene procedures within 12-18 hours prior to each visit.
* Refrain from eating, drinking or smoking for four hours prior to each visit.

Exclusion Criteria:

* Lip, tongue, or other form of oral piercing.
* Fixed or removable orthodontic appliance (such as bridges, braces or dentures).
* Pregnancy or breast-feeding at any time during the trial.
* Any medical, dental or psychiatric condition, abnormality or history, or use of any product or drug, that (per protocol or in the opinion of the investigator) may increase the risk to the subject associated with trial participation or investigational product administration, or interfere with the interpretation of trial results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2011-12-02 (Actual); Study Completion 2011-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Araujo, DDS, MS, PhD, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (1):
- BioSci Research Inc., Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5% Hydroalcohol Mouthrinse | 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse
Started | 44 | 43
Completed | 43 | 43
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5% Hydroalcohol Mouthrinse | 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (10.35) | 34.0 (8.05) | 34.8 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 53
  Male | 21 | 13 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 39 | 37 | 76
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 4 | 4 | 8
  Black or African American | 14 | 9 | 23
  White | 23 | 26 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Smoker [Count of Participants; unit: Participants] — Number of participants who smoke
  Participants
    Yes | 4 | 6 | 10
    No | 40 | 37 | 77
Smokeless Tabacco Use [Count of Participants; unit: Participants] — Number of Participants who use smokeless tobacco
  Participants
    Yes | 1 | 0 | 1
    No | 43 | 43 | 86
Mean Plaque Index - Whole Mouth [Mean (Standard Deviation); unit: Units on a scale] — Plaque was assessed on a scale of 0-5 using the Turesky modification of the Quigley-Hein Plaque Index, where 0=No plaque and 5=Plaque covering 2/3 or more of surface.
  Units on a scale | 2.996 (0.2222) | 2.926 (0.2866) | 2.961 (0.257)
Modified Gingival Index - Whole Mouth [Mean (Standard Deviation); unit: Units on a scale] — Gingivitis was assessed by scoring inflammation on a 0-4 scale, according to the Modified Gingival Index (MGI) where 0=Normal and 4=Severe Inflammation
  Units on a scale | 2.196 (0.0989) | 2.172 (0.1132) | 2.184 (0.106)
Gingival Bleeding Index - Whole Mouth [Mean (Standard Deviation); unit: Units on a scale] — Bleeding after periodontal probe was assessed by scores on a scale of 0-2 using the Gingival Bleeding Index (BI), where 0=Absence of Bleeding after 30 Seconds and 2=Immediate Bleeding.
  Units on a scale | 0.137 (0.0614) | 0.129 (0.0634) | 0.133 (0.062)
Microbiological Assessments - Absolute Counts [Mean (Standard Deviation); unit: 10^5 bacterial cells] — A checkerboard DNA-DNA hybridization was conducted to estimate the # of bacterial cells in plaque samples. DNA from lysed bacteria cells was detected using fluorescent probes for different bacterial species. The sensitivity of the assay was 10^4 cells; failure to detect a signal was recorded as 0. Signals were converted to absolute counts by comparison with fluorescent signals of standards of known concentrations. The following hybridized categories of bacteria were analyzed: Actinomyces species, Purple complex, Yellow complex, Green complex, Orange complex, Red complex, & Other species
  10^5 bacterial cells
    Actinomyces species | 3.206 (1.7377) | 3.319 (1.8306) | 3.262 (1.7747)
    Purple complex | 2.207 (1.7989) | 2.181 (1.888) | 2.194 (1.5193)
    Yellow complex | 2.400 (2.2929) | 2.535 (1.5893) | 2.467 (1.9664)
    Green complex | 7.988 (8.8495) | 6.841 (6.5277) | 7.421 (7.7653)
    Orange complex | 5.252 (3.6072) | 4.923 (3.6457) | 5.089 (3.6089)
    Red complex | 1.638 (0.8182) | 1.509 (0.8192) | 1.574 (0.8165)
    Other species | 7.646 (6.1549) | 7.322 (6.2088) | 7.486 (6.1477)
Microbiological Assessments - LOG Counts [Mean (Standard Deviation); unit: LOG counts of bacterial cells] — A checkerboard DNA-DNA hybridization was conducted to estimate the # of bacterial cells in plaque samples. DNA from lysed bacteria cells was detected using fluorescent probes for different bacterial species. The sensitivity of the assay was 10^4 cells; failure to detect a signal was recorded as 0. Signals were converted to log counts by comparison with fluorescent signals of standards of known concentrations. The following hybridized categories of bacteria were analyzed: Actinomyces species, Purple complex, Yellow complex, Green complex, Orange complex, Red complex, & Other species
  LOG counts of bacterial cells
    Actinomyces species | 5.410 (0.3647) | 5.440 (0.2935) | 5.425 (0.3298)
    Purple complex | 5.213 (0.3985) | 5.255 (0.3107) | 5.234 (0.3563)
    Yellow complex | 5.249 (0.3433) | 5.302 (0.3284) | 5.275 (0.3351)
    Green complex | 5.717 (0.4232) | 5.660 (0.4038) | 5.689 (0.4123)
    Orange complex | 5.603 (0.3506) | 5.583 (0.3226) | 5.593 (0.3352)
    Red complex | 5.149 (0.2624) | 5.110 (0.2584) | 5.130 (0.2596)
    Other species | 5.756 (0.3524) | 5.722 (0.3660) | 5.739 (0.3575)

OUTCOME MEASURES:

1. Primary Outcome: Whole-mouth Mean Modified Gingival Index (MGI)
Description: Gingivitis was assessed by scoring inflammation on a 0-4 scale, according to the Modified Gingival Index (MGI) where 0=Normal and 4=Severe Inflammation.
Time Frame: 4 weeks
Population: Intent to treat population was analyzed; one subject discontinued from the study prior to Week 4.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 5% Hydroalcohol Mouthrinse | 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse
Number analyzed (Participants) | 43 | 43
Units on a scale | 2.199 (0.0934) | 1.948 (0.1548)
Statistical Analysis 1: Comparison: 5% Hydroalcohol Mouthrinse vs 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse; Test type: Superiority — The null hypothesis was the Week 4 mean is equal between the two cells. The alternative hypothesis was the Week 4 mean is not equal between the two cells; p < 0.001, ANCOVA; Terms for treatment as a factor & baseline as a covariate; Mean Difference (Net) = -0.234, 95% CI 2-sided [-0.276 to -0.192], Standard Error of Mean 0.0211

2. Primary Outcome: Whole-mouth Mean Plaque Index (PI)
Description: Plaque was assessed on a scale of 0-5 using the Turesky modification of the Quigley-Hein Plaque Index, where 0=No plaque and 5=Plaque covering 2/3 or more of surface.
Time Frame: 4 weeks
Population: Intent to treat population was analyzed; one subject discontinued from the study prior to Week 4.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 5% Hydroalcohol Mouthrinse | 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse
Number analyzed (Participants) | 43 | 43
Units on a scale | 2.922 (0.1953) | 1.634 (0.5724)
Statistical Analysis 1: Comparison: 5% Hydroalcohol Mouthrinse vs 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA; Terms for treatment as a factor & baseline as a covariate; Mean Difference (Net) = -1.232, 95% CI 2-sided [-1.392 to -1.071], Standard Error of Mean 0.0806

3. Secondary Outcome: Whole-mouth Mean Modified Gingival Index (MGI)
Description: Gingivitis was assessed by scoring inflammation on a 0-4 scale, according to the Modified Gingival Index, where 0=Normal and 4=Severe Inflammation.
Time Frame: 2 weeks
Population: Intent to treat population was used for analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 5% Hydroalcohol Mouthrinse | 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse
Number analyzed (Participants) | 44 | 43
Units on a scale | 2.189 (0.1014) | 2.067 (0.1185)
Statistical Analysis 1: Comparison: 5% Hydroalcohol Mouthrinse vs 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse; Test type: Superiority — The null hypothesis was the Week 2 mean is equal between the two cells. The alternative hypothesis was the Week 2 mean is not equal between the two cells; p < 0.001, ANCOVA; Terms for treatment as a factor & baseline as a covariate; Mean Difference (Net) = -0.106, 95% CI 2-sided [-0.140 to -0.071], Standard Error of Mean 0.0173

4. Secondary Outcome: Whole-mouth Mean Plaque Index (PI)
Description: as for outcome 2
Time Frame: 2 Weeks
Population: The intent-to-treat population was used for analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 5% Hydroalcohol Mouthrinse | 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse
Number analyzed (Participants) | 44 | 43
Units on a scale | 2.880 (0.2678) | 1.987 (0.6539)
Statistical Analysis 1: Comparison: 5% Hydroalcohol Mouthrinse vs 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.001, ANCOVA; Terms for treatment as a factor & baseline as a covariate; Mean Difference (Net) = -0.830, 95% CI 2-sided [-1.020 to -0.639], Standard Error of Mean 0.0957

5. Secondary Outcome: Whole-mouth Mean Bleeding Index (BI)
Description: Bleeding after periodontal probe was assessed by scores on a scale of 0-2 using the Gingival Bleeding Index (BI), where 0=Absence of Bleeding after 30 Seconds and 2=Immediate Bleeding.
Time Frame: 2 Weeks
Population: Intent to treat population was analyzed.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 5% Hydroalcohol Mouthrinse | 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse
Number analyzed (Participants) | 44 | 43
Units on a scale | 0.123 (0.0569) | 0.074 (0.0528)
Statistical Analysis 1: Comparison: 5% Hydroalcohol Mouthrinse vs 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.001, ANCOVA; Terms for treatment as a factor & baseline as a covariate; Mean Difference (Net) = -0.044, 95% CI 2-sided [-0.059 to -0.029], Standard Error of Mean 0.0076

6. Secondary Outcome: Whole-mouth Mean Bleeding Index (BI)
Description: as for outcome 5
Time Frame: 4 Weeks
Population: Intent to treat population was analyzed; one subject discontinued from the study prior to Week 4.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 5% Hydroalcohol Mouthrinse | 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse
Number analyzed (Participants) | 43 | 43
Units on a scale | 0.120 (0.0524) | 0.057 (0.0520)
Statistical Analysis 1: Comparison: 5% Hydroalcohol Mouthrinse vs 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA; Terms for treatment as a factor & baseline as a covariate; Mean Difference (Net) = -0.060, 95% CI 2-sided [-0.078 to -0.043], Standard Error of Mean 0.0087

7. Secondary Outcome: Microbiological Assessments - Absolute Counts
Description: An assay (a checkerboard DNA-DNA hybridization) was conducted to estimate the number of bacterial cells in collected plaque samples. First, the bacterial cells were lysed (split open) in solution. DNA from the bacteria was then detected using fluorescent probes for different bacterial species. The sensitivity of the assay was 10^4 cells and failure to detect a signal was recorded as zero. Signals were converted to absolute counts by comparison with the fluorescent signal of standards of known concentrations.
  The following hybridized categories of bacteria were analyzed:
  * Actinomyces species
  * Purple complex
  * Yellow complex
  * Green complex
  * Orange complex
  * Red complex
  * Other species
Time Frame: 4 weeks
Population: Intent to treat population was analyzed; one subject discontinued from the study prior to Week 4.
Measure: Mean (Standard Deviation); unit: 10^5 bacterial cells
Arm/Group | 5% Hydroalcohol Mouthrinse | 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse
Number analyzed (Participants) | 43 | 43
10^5 bacterial cells
  Actinomyces species | 1.868 (1.5514) | 1.847 (1.2609)
  Purple complex | 0.910 (0.9723) | 0.663 (0.6454)
  Yellow complex | 1.050 (0.8595) | 1.018 (0.7001)
  Green complex | 4.530 (3.8225) | 3.174 (2.4853)
  Orange complex | 3.562 (3.1562) | 3.602 (2.4298)
  Red complex | 1.346 (1.0472) | 1.111 (0.6017)
  Other Species | 4.471 (3.9108) | 3.385 (2.3474)

8. Secondary Outcome: Microbiological Assessments - LOG Counts
Description: An assay (a checkerboard DNA-DNA hybridization) was conducted to estimate the number of bacterial cells in collected plaque samples. First, the bacterial cells were lysed (split open) in solution. DNA from the bacteria was then detected using fluorescent probes for different bacterial species. The sensitivity of the assay was 10^4 cells and failure to detect a signal was recorded as zero. Signals were converted to log counts by comparison with the fluorescent signal of standards of known concentrations.
  The following hybridized categories of bacteria were analyzed:
  * Actinomyces species
  * Purple complex
  * Yellow complex
  * Green complex
  * Orange complex
  * Red complex
  * Other species
Time Frame: 4 weeks
Population: Intent to treat population was analyzed; one subject discontinued from the study prior to Week 4.
Measure: Mean (Standard Deviation); unit: LOG counts of bacterial cells
Arm/Group | 5% Hydroalcohol Mouthrinse | 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse
Number analyzed (Participants) | 43 | 43
LOG counts of bacterial cells
  Actinomyces species | 5.089 (0.4432) | 5.154 (0.3491)
  Purple complex | 4.721 (0.5443) | 4.617 (0.4546)
  Yellow complex | 4.882 (0.3674) | 4.915 (0.2855)
  Green complex | 5.477 (0.4354) | 5.400 (0.2935)
  Orange complex | 5.401 (0.3761) | 5.461 (0.3008)
  Red complex | 5.012 (0.3354) | 4.977 (0.2637)
  Other Species | 5.509 (0.3637) | 5.433 (0.3005)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of informed consent through subject's last study procedure (Week 4, unless terminated early). Serious adverse events (SAE) reported to the site were also reportable within 30 calendar days of last procedure/visit and longer if considered study-related; there was no specific cut-off date for this reporting,
Arm/Group | 5% Hydroalcohol Mouthrinse | 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/43
Other Adverse Events (participants affected / at risk) | 0/44 | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5% Hydroalcohol Mouthrinse (N=44) | 0.15% Ethyl Lauroyl Arginate HCl-containing Mouthrinse (N=43)
Testicular Swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must provide Sponsor 60 days to review any publication (unless expedited review requested); if includes Sponsor's confidential info, written Sponsor approval is required. Sponsor may require another 60 days' delay to file patent app. If multicenter, PI agrees 1st publication is joint publication. If join publication not submitted within 24 months of study end or Sponsor confirms there will be no joint publication, PI may publish the results individually following previous guidelines.